CLINICAL TRIAL: NCT07377851
Title: Erythrocyte Carbonic Anhydrase II as a Marker of Metabolic Adaptation to Basketball-Specific High-Intensity Interval Training
Brief Title: Carbonic Anhydrase II Responses to Basketball-Specific High-Intensity Interval Training
Acronym: CAII-BASKET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Recep Soslu, Associate Professor, Karamanoğlu Mehmetbey University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 03-2023/02
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Metabolic Adaptation to High-Intensity Interval Training
Keywords: Carbonic Anhydrase II; Exercise Physiology; Metabolic Adaptation; High-Intensity Interval Training; Basketball Training

STUDY DESIGN:
Masking Description: No additional parties were masked. The study was conducted as an open-label trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Basketball-Specific High-Intensity Interval Training (Experimental): Participants completed a basketball-specific high-intensity interval training program designed to induce metabolic adaptations. All participants were assigned to this single intervention arm and completed the same training protocol.
  Interventions: Behavioral: Basketball-Specific High-Intensity Interval Training

INTERVENTIONS:
Behavioral: Basketball-Specific High-Intensity Interval Training — A structured basketball-specific high-intensity interval training program consisting of repeated bouts of intense exercise interspersed with short recovery periods, designed to induce metabolic adaptations.

SUMMARY:
This study aims to examine whether erythrocyte carbonic anhydrase II can be used as a biological marker of metabolic adaptation to basketball-specific high-intensity interval training. Carbonic anhydrase II is an enzyme involved in acid-base balance and carbon dioxide transport, and it may reflect physiological adaptations to intense exercise.

Healthy basketball players participated in a structured high-intensity interval training program designed to reflect the physical demands of basketball. Blood samples and performance-related measurements were collected before and after the training period to evaluate changes in erythrocyte carbonic anhydrase II levels and related metabolic responses.

The findings of this study are expected to improve the understanding of exercise-induced metabolic adaptations and to explore the potential use of erythrocyte carbonic anhydrase II as a practical biomarker for monitoring training responses in basketball players.

DETAILED DESCRIPTION:
This study was designed to investigate erythrocyte carbonic anhydrase II as a potential biomarker of metabolic adaptation to basketball-specific high-intensity interval training. Carbonic anhydrase II plays a key role in acid-base regulation and carbon dioxide transport, which are critical physiological processes during repeated high-intensity exercise.

Participants were healthy basketball players who completed a structured high-intensity interval training program reflecting the intermittent and high-demand nature of basketball activity. The training protocol consisted of repeated bouts of intense exercise interspersed with short recovery periods, consistent with established basketball-specific conditioning practices.

Blood samples were obtained at predefined time points to assess erythrocyte carbonic anhydrase II levels. These biochemical measurements were evaluated alongside selected performance and physiological indicators to characterize training-induced metabolic adaptations. All assessments were conducted under standardized conditions to minimize variability related to diet, hydration, and recent physical activity.

The study followed an observational pre-post design without clinical intervention beyond the prescribed training program. No experimental drugs or medical devices were used. Safety monitoring was conducted throughout the study period, and no serious adverse events were anticipated given the low-risk nature of the exercise protocol and the healthy status of the participants.

This study seeks to contribute to the growing body of research on exercise-related biomarkers by examining whether erythrocyte carbonic anhydrase II may provide practical insight into metabolic adaptation to sport-specific high-intensity training.

ELIGIBILITY:
Inclusion Criteria:

Healthy male and female basketball players aged 18 years or older

Actively participating in regular basketball training at the time of the study

Free from known cardiovascular, metabolic, or respiratory diseases

No musculoskeletal injury that could limit participation in high-intensity exercise

Willingness to participate in a basketball-specific high-intensity interval training program

Ability to provide written informed consent

Exclusion Criteria:

Presence of any diagnosed cardiovascular, metabolic, or respiratory disease

Use of medications or supplements known to affect metabolic or acid-base balance

Acute or chronic musculoskeletal injury within the previous three months

Participation in another structured training or research intervention during the study period

Failure to comply with the training protocol or assessment procedures

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-01-10 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Erythrocyte Carbonic Anhydrase II Levels | Baseline( week 0) and post training (week 8)
  The primary outcome is the change in erythrocyte carbonic anhydrase II levels measured before and after the basketball-specific high-intensity interval training program. Erythrocyte carbonic anhydrase II was assessed from blood samples as an indicator of metabolic adaptation to high-intensity exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Karamanoğlu Mehmetbey University, Faculty of Sport Sciences, Karaman, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No